CLINICAL TRIAL: NCT07001527
Title: Dressing Impregnated With Chlorhexidine and Vancomycin for the Prophylaxis of Central Venous Catheter-related Infections - a Randomized Trial
Acronym: Dressing RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Evangelico de Curitiba (Other)
Responsible Party: Principal Investigator, Felipe Francisco Bondan Tuon, Professor, Pontifícia Universidade Católica do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PUCPR-Dressing; 0001 (Other Grant/Funding Number: Researcher)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chlorhexidine
Keywords: chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impregnated (Active Comparator): Impregnated
  Interventions: Device: Chlorhexidine
- Control (Placebo Comparator): COmmon dressing
  Interventions: Device: Chlorhexidine

INTERVENTIONS:
Device: Chlorhexidine — dressing impregnated
  Other Names: Impregnated dressing
Device: Chlorhexidine — COmmon dressing
  Other Names: COmmon dressing

SUMMARY:
You are being invited as a volunteer to participate in the study "Dressing impregnated with chlorhexidine and vancomycin for the prophylaxis of central venous catheter-related infections." The objective is to evaluate the incidence of bloodstream infection related to the catheter in ICU patients with central venous catheters (CVC), using dressings impregnated or not with chlorhexidine/vancomycin. We believe this study is important as it aims to evaluate a new dressing method intended to reduce bloodstream-related infections.

ELIGIBILITY:
IInclusion criteria included: age over 18 years, admitted to the ICU, need for a CVC placed in the ICU by the trained team, use of the CVC for a period exceeding 72 hours, and intact skin in the area of contact with the dressing. CVC inserted outside the ICU and need for two CVCs in the same patient simultaneously were exclusion criteria. A subsequent CVC could not be randomized. Other infections were not excluded during the evaluation. Only short-term CVC were evaluated (long-term and hemodialysis were excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Infection | 30 days
  CRBSI was the primary endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- PUCPR, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No